CLINICAL TRIAL: NCT02948166
Title: Prospective Randomized Clinical Trial of the Remote Endarterectomy and the Femoral Arteries Endovascular Treatments in Patients With the Femoral Artery Occlusive Disease (TASC C, D)
Brief Title: Remote Endarterectomy and Endovascular Treatments in Patients With the Femoral Artery Occlusive Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: N-RICP-468
Record Dates: First submitted 2016-09-25; First posted 2016-10-28 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Steno-occlusive Desease of Femoro-popliteal Arterial Segment
Keywords: remote endarterectomy; Angioplasty with stenting of the superficial femoral artery
MeSH Terms: interventions — Angioplasty; Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stenting of the femoral artery (Active Comparator): A standard endovascular treatment of the steno-occlusive lesion in femoro-popliteal arterial segment.
  Interventions: Procedure: Angioplasty with stenting of the femoral artery
- Open surgery (Experimental): Performed open endarterectomy of the common, deep, initial of superficial femoral artery. Delamination factory complex into the lumen of the loop. After that, the translational and rotational motions loops under fluoroscopic guidance, continuing detachment of plaque in the antegrade direction to the distal end of plaque. Plastic arteriotomnyh wounds performed patches of ksenoperikard treated with epoxy compounds. Control patency of the arterial bed is performed intraoperatively by X-ray angiography.
  Interventions: Procedure: Open surgery

INTERVENTIONS:
Procedure: Angioplasty with stenting of the femoral artery — A standard endovascular exposure is carried out under local anesthesia and a lesioned arterial segment is visualized. Stenosis or artery occlusion is passed by the hydrophilic guide. During the occlusion transluminal or subintimal artery recanalization (most frequently mixed) is conduced. Then balloon angioplasty of stenosis or occlusion are carried out. After the angiographic control if necessary stent (balloon expandable or self-expanding) of all the extension is mounted.
  Arms: Stenting of the femoral artery
Procedure: Open surgery — Performed open endarterectomy of the common, deep, initial of superficial femoral artery. Proximal plaque exfoliate as far as possible in the superficial femoral artery. After that, the translational and rotational motions loops under fluoroscopic guidance, continuing detachment of plaque in the antegrade direction to the distal end of plaque. Plastic of arteriotomy wounds performed patches of ksenoperikard treated with epoxy compounds. Control patency of the arterial vessel is performed intraoperatively by X-ray angiography. When rendering residual stenosis or intimal dissection, limiting blood flow, complemented by endovascular intervention plasticity.
  Arms: Open surgery

SUMMARY:
Comparison of two methods for revascularization of the superficial femoral artery: remote endarterectomy vs. stenting of the superficial femoral artery cin patients with steno-occlusive lesion of the femoro-popliteal segment of TASC C, D

DETAILED DESCRIPTION:
Reported local percutaneous angioplasty and stenosis of femoral popliteal arteries indicate that the primary technical and clinical success above 95%. The technical success of recanalization of long occlusions femoral arteries less than 80%. Improvement of endovascular equipment designed for the treatment of total occlusions, increases the technical success of recanalization. The materials of the TASC II summarizes the results of several large studies that presented data on the operated segment artery patency at 56-73,7% within 2 years of observation. An alternative method of revascularization own femoral artery is remote endarterectomy. The two-year primary patency at remote endarterectomy is 86% (Moll F.L., Iio G.H. Closed superficial femoral artery endarterectomy: a 2-year follow up. Cardiovasc Surg. 1997; 5: 398-400). Primary assisted patency for 33 months 88% (Rosenthal D, Martin JD, Schubart PJ, Wellons ED. Remote. superﬁcial femoral artery endarterectomy. J Cardiovasc Surg. (Torino) 2004; 45: 185-192). The length of the occlusion is not a limitation to the use of remote endarterectomy. Primary patency at 31 months was 60%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with occlusive lesions of C and D type femoral artery and with chronic lower limb ischemia (II-IV degree by Fontaine, 4-6 degree by Rutherford)
* Patients who consented to participate in this study.

Exclusion Criteria:

* Chronic heart failure of III-IV functional class by NYHA classification.
* Decompensated chronic "pulmonary" heart
* Severe hepatic or renal failure (bilirubin> 35 mmol / l, glomerular filtration rate <60 mL / min);
* Polyvalent drug allergy
* Cancer in the terminal stage with a life expectancy less than 6 months;
* Acute ischemic
* Expressed aortic calcification tolerant to angioplasty
* Patients with significant common femoral artery lesion
* Patient refusal to participate or continue to participate in the study

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
the change of lumen in target vessel | Baseline, 3 days after the operation, 6 month, 12 month, 2, 3 years

SECONDARY OUTCOMES:
Number of participants with a successful procedure of revascularization. | During the operation.
Number of participants with complications during the operation. | During the operation.
Number of participants with limb salvage | Baseline, 3 days after the operation, 6 month, 12 month, 2, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Karpenko, Study Director — cientific-Research Institute of Circulation Pathology named after Academician E. Meshalkin
Locations (1):
- Federal State Institution Academician E.N.Meshalkin Novosibirsk State Research Institute Of Circulation Pathology Rusmedtechnology, Novosibirsk, Russia